CLINICAL TRIAL: NCT06834685
Title: Evaluating Laser Photobiomodulation for the Treatment of Neuropathic Pain in Chemotherapy-induced Peripheral Neuropathy: a Randomized, Non-comparative, Placebo-controlled, Single-blinded, Phase II Clinical Trial in Cancer Patients
Brief Title: Evaluating Laser Photobiomodulation for the Treatment of Neuropathic Pain in Chemotherapy-induced Peripheral Neuropathy in Cancer Patients
Acronym: NEUROdoux
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PROICM 2024605 NEU; 2024-A02524-43 (Other: ID-RCB)
Record Dates: First submitted 2025-02-07; First posted 2025-02-19 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Cancer Survivors; Peripheral Neuropathic Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (Experimental): Photobiomodulation sessions (2 per week for 4 weeks, 8 sessions in total) will be delivered by certified laser safety clinicians (i.e., algologists, pain nurses or neuropsychologists).
  The treatment will be administered by an ATP38 device delivering a power of 4 Joules/cm2 at wavelengths of 620 and 820 nm. The light will be applied to all hands and/or feet for 13 minutes. The order of transfer between feet and hands will be counterbalanced so that, half of the sessions will have started with feet, and the other half will have started with hands. The dose will be specified at each session.
  Patients will be treated in a sitting position (to treat the hands) or a semi-seated position (for feet). They will wear opaque glasses to ensure the safety of the laser and the blind condition of treatment
  Interventions: Device: Photobiomodulation sessions
- Control arm (No Intervention): In the sham therapy, patients will have the same procedure as the laser intervention (i.e., visit schedule, eye mask, equipment, and application body regions), but without joules.
  Patients in this placebo arm will have the opportunity to receive the real treatment at the end of the study if they wish.

INTERVENTIONS:
Device: Photobiomodulation sessions — The treatment will be administered by an ATP38 device delivering a power of 4 Joules/cm2 at wavelengths of 620 and 820 nm
  Arms: Experimental arm

SUMMARY:
Chemotherapy-induced peripheral neuropathy (CIPN) (including taxanes, platinum, al pervenche from Madagascar alkaloids...), is a frequent secondary effect of treatments: 68% at 1-month post-chemotherapy, 60% at 3 months and 30% after 6 months. Symptoms associated with CIPN are usually symmetric and bilateral (typical distribution in "gloves and socks") inducing sensory alterations, paresthesias, dysesthesias, numbness and pain. Neuropathic Pain (NP) is an important characteristic of CIPN, affects 25-80% of patients with CIPN, and reduces quality of life (e.g., concomitant psychological distress, risks of falls, risks of neurocognitive impairments, and sleep disorders).

In severe cases, it is even necessary to delay and/or reduce the dose of chemotherapy. The benefit of drug interventions on NP remains limited. To date, there are no proven preventive strategies and few evidence-based treatment options for CIPN. Also, the use of complementary or non-pharmacological interventions are common, including photobiomodulation (PBM).

PBM is the therapeutic use of non-ionizing laser light for its anti-inflammatory and regenerative effects. Its use is currently recommended only for the prevention of oral mucositis related to cancer treatments. Recent preliminary clinical evidence suggests that PBM may be beneficial to established CIPN, with safety and improvement beyond the intervention. However, to date, clinical trials are rare, have methodological weaknesses, and/or focus on global CIPN. The overall objectives of the study are therefore to assess the effectiveness, feasibility and safety of the PBM for treating NP in the CIPN.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 years minimum;
* Patient treated at the Montpellier Cancer Institute for a cancer (whatever the location) requiring a chemotherapy;
* Patient with significant NP defined as a score of 4 at the clinician-rated DN4 ;
* Patient with a NP for at least 3 months after the end of an adjuvant or neo-adjuvant chemotherapy;
* Women of childbearing potential must have a pregnancy urinary test within a maximum of 7 days before starting the study treatment. A negative result must be documented before study treatment is started. Women without reproductive potential are postmenopausal women or women who have undergone permanent sterilisation (e.g. tubal occlusion, hysterectomy, bilateral salpingectomy);
* Effective contraception for women of childbearing age
* Patient having signed informed consent prior to any study procedure;
* Patient affiliated to a French social protection system;
* Patient sufficiently fluent in French to complete questionnaires, as the investigator clinical discretion.

Exclusion Criteria:

* Patient unable to come twice a week to the Montpellier Cancer Institute;
* Patient unable to sit for a 30-minutes period;
* Patient with an open wound or ulcer on the treatment area;
* Patient whose diagnosis of peripheral neuropathy is due to another cause (n.b., diabetes without neuropathy will not be a specific exclusion);
* Patient with uncontrolled psychiatric illness or neurocognitive impairment that may interfere with assessments, as the investigator clinical discretion;
* Patient whose estimated life expectancy is less than 3 months, as estimated by a clinical investigator;
* Patient using another concurrent non-pharmacological intervention or complementary therapy for neuropathy during the study;
* Patient who has been treated with CAPSAISINE during the previous 3 months;
* Patient with pacemaker;
* Epileptic patient;
* Patient with photosensitive medications, or any medical condition causing sensitivity to light (n.b., Lupus);
* Pregnant and/or breastfeeding woman;
* Patient with primary tumor and/or metastases in areas to be treated by BPM (i.e., hands and/or feet);
* Patient with pre-existing eye disease (such as maculopathy, glaucoma, cataract and retinal lesions), or a history of family eye diseases;
* Patient who has been already been treated with photobiomodulation on the area of interest.
* Participation in another concomitant clinical study with neuropathic pain or chemo-induced peripheral neuropathy as the primary endpoint.
* Presence of a tattoo on the area to be treated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-10-07 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the efficacy of photobiomodulation on neuropathic pain in a experimental group and evaluate the placebo effect in a controlled group | from the baseline to 12 weeks after the treatment
  the proportion of responders to a photobiomodulation intervention on their neuropathic pain at 12 weeks

SECONDARY OUTCOMES:
Description of the evolution of neuropathic pain | from the baseline to 6 months after the treatment
  description by the scores of the clinician-rated neuropathic pain questionnaire (from 0 to 10, 0 no neuropathic pain, 10 : worst neuropatic pain)
Description of the evolution of neuropathic pain | from the baseline to 6 months after the treatment
  description by the scores of the self-questionnaire Neuropathic Pain Symptom Inventory (from 0 to 100, 0 no neuropathic pain, 100 : worst neuropatic pain)
Exploration of the evolution of global pain measures | from the baseline to 6 months after the treatment
  The global pain will be assessed using the scores of the self-questionnaire Brief Pain Inventory (from 0 to 110, 0 no neuropathic pain, 110 : worst neuropatic pain)
Exploration of the evolution of global pain measures | from the baseline to 6 months after the treatment
  The global pain will be assessed using the scores of the Numeric Scale of pain (from 0 to 10, 0 no pain, 10 worst pain)
Description of the evolution of the Chemotherapy-induced peripheral neuropathy | from the baseline to 6 months after the treatment
  The chemotherapy-induced peripheral neuropathy will be described using the scores of the self-questionnaire FACT/GOG-Ntx-13, and the grade of chemotherapy-induced peripheral neuropathy assessed by the clinician via the Common Terminology Criteria for Adverse Events (ranging from 0 to 5, a high score indicates a strong neuropathy).
Exploration of the evolution of quality of life | from the baseline to 6 months after the treatment
  The quality of life will be explored using the self-questionnaire Functional Assessment of Chronic illness Therapy-Global scores [the global score and its 4 sub-scales scores (physical, social/family, emotional, functional] and the number of falls reported by the patient during the last month (from 0 to 108, 0 bad quality of life, 108 good quality of life)
Exploration of the evolution of sleep disorders | from the baseline to 6 months after the treatment
  Sleep disorders will be explored using the self-assessment Sleep Severity Index (ISI).
Description of the evolution of neurocognitive executive functioning | from the baseline to 6 months after the treatment
  Neurocognitive functioning will be assessed using the clinician-rated scores of the test modified-Delis-Kaplan Executive Function System (m-DKEFS)
Description of the evolution of neurocognitive executive functioning | from the baseline to 6 months after the treatment
  Neurocognitive functioning will be assessed using the scores of the Trail Making Test (TMT A and B)
Assessment of the photobiomodulation adherence | from the baseline to 4 weeks after the beginning of the treatment
  The adherence to the intervention will be assessed by the number of PBM sessions performed by patients
Evaluation of the safety of the photobiomodulation | from the baseline to 6 months after the treatment
  The safety of PBM will be assessed by the number and the severity of target adverse events recorded during the study period, using the CTCAE scale (v5.0)
Assessment of emotional distress | from the baseline to 4 weeks after the treatment
  Emotional distress will be measured by the score of the Hospital Anxiety and Depression Scale (HADS) Questionnaire at baseline and at the end of photobiomodulation treatment

CONTACTS AND LOCATIONS:
Overall Officials: Estelle GUERDOUX, PHD, Study Director — INSTITUT REGIONAL DU CANCER DE MONTPELLIER
Locations (1):
- ICM, Montpellier, France

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared at an individual level. Those data will be part of the study database including all enrolled patients All participant data collected during the trial, after encoding with an inclusion number, 1st letter of the name and surname may be shared.
  The data of the participants will be available upon request and with the completion of a contract between the promoter and the applicant.
  The study protocol, the statistical analysis plan (PAS) and the analytical code may also be subject to data sharing as part of a transfer contract (RGPD)

REFERENCES:
- [Background] Seretny M, Currie GL, Sena ES, Ramnarine S, Grant R, MacLeod MR, Colvin LA, Fallon M. Incidence, prevalence, and predictors of chemotherapy-induced peripheral neuropathy: A systematic review and meta-analysis. Pain. 2014 Dec;155(12):2461-2470. doi: 10.1016/j.pain.2014.09.020. Epub 2014 Sep 23. PMID 25261162
- [Background] Joy L, Jolien R, Marithe C, Stijn E, Laura S, Hilde L, Sandra B, Wendy N, Ruth H, Liesbeth R, Sylvana S, Sylvia H, Jeroen M. The use of photobiomodulation therapy for the prevention of chemotherapy-induced peripheral neuropathy: a randomized, placebo-controlled pilot trial (NEUROLASER trial). Support Care Cancer. 2022 Jun;30(6):5509-5517. doi: 10.1007/s00520-022-06975-x. Epub 2022 Mar 21. PMID 35312857
- [Background] Teng C, Egger S, Blinman PL, Vardy JL. Evaluating laser photobiomodulation for chemotherapy-induced peripheral neuropathy: a randomised phase II trial. Support Care Cancer. 2022 Dec 17;31(1):52. doi: 10.1007/s00520-022-07463-y. PMID 36526802
- [Background] Zadik Y, Arany PR, Fregnani ER, Bossi P, Antunes HS, Bensadoun RJ, Gueiros LA, Majorana A, Nair RG, Ranna V, Tissing WJE, Vaddi A, Lubart R, Migliorati CA, Lalla RV, Cheng KKF, Elad S; Mucositis Study Group of the Multinational Association of Supportive Care in Cancer/International Society of Oral Oncology (MASCC/ISOO). Systematic review of photobiomodulation for the management of oral mucositis in cancer patients and clinical practice guidelines. Support Care Cancer. 2019 Oct;27(10):3969-3983. doi: 10.1007/s00520-019-04890-2. Epub 2019 Jul 8. PMID 31286228
- [Background] Escritt K, Mann M, Nelson A, Harrop E. Hope and meaning-making in phase 1 oncology trials: a systematic review and thematic synthesis of qualitative evidence on patient-participant experiences. Trials. 2022 May 16;23(1):409. doi: 10.1186/s13063-022-06306-9. PMID 35578308
- [Background] D'Souza RS, Alvarez GAM, Dombovy-Johnson M, Eller J, Abd-Elsayed A. Evidence-Based Treatment of Pain in Chemotherapy-Induced Peripheral Neuropathy. Curr Pain Headache Rep. 2023 May;27(5):99-116. doi: 10.1007/s11916-023-01107-4. Epub 2023 Apr 14. PMID 37058254
- [Background] Molinares D, Kurtevski S, Zhu Y. Chemotherapy-Induced Peripheral Neuropathy: Diagnosis, Agents, General Clinical Presentation, and Treatments. Curr Oncol Rep. 2023 Nov;25(11):1227-1235. doi: 10.1007/s11912-023-01449-7. Epub 2023 Sep 13. PMID 37702983
- [Background] Kerckhove N, Collin A, Conde S, Chaleteix C, Pezet D, Balayssac D, Guastella V. [Chemotherapy-induced peripheral neuropathy: Symptomatology and epidemiology]. Bull Cancer. 2018 Nov;105(11):1020-1032. doi: 10.1016/j.bulcan.2018.07.009. Epub 2018 Sep 20. French. PMID 30244980
- [Background] Rao V, Bhushan R, Kumari P, Cheruku SP, Ravichandiran V, Kumar N. Chemobrain: A review on mechanistic insight, targets and treatments. Adv Cancer Res. 2022;155:29-76. doi: 10.1016/bs.acr.2022.04.001. Epub 2022 May 11. PMID 35779876
- [Background] Ong WY, Stohler CS, Herr DR. Role of the Prefrontal Cortex in Pain Processing. Mol Neurobiol. 2019 Feb;56(2):1137-1166. doi: 10.1007/s12035-018-1130-9. Epub 2018 Jun 6. PMID 29876878
- [Background] McCrary JM, Goldstein D, Trinh T, Timmins HC, Li T, Menant J, Friedlander M, Lewis CR, Hertzberg M, O'Neill S, King T, Bosco A, Harrison M, Park SB. Balance Deficits and Functional Disability in Cancer Survivors Exposed to Neurotoxic Cancer Treatments. J Natl Compr Canc Netw. 2019 Aug 1;17(8):949-955. doi: 10.6004/jnccn.2019.7290. PMID 31390588
- [Background] Winters-Stone KM, Horak F, Jacobs PG, Trubowitz P, Dieckmann NF, Stoyles S, Faithfull S. Falls, Functioning, and Disability Among Women With Persistent Symptoms of Chemotherapy-Induced Peripheral Neuropathy. J Clin Oncol. 2017 Aug 10;35(23):2604-2612. doi: 10.1200/JCO.2016.71.3552. Epub 2017 Jun 6. PMID 28586243
- [Background] Hong JS, Tian J, Wu LH. The influence of chemotherapy-induced neurotoxicity on psychological distress and sleep disturbance in cancer patients. Curr Oncol. 2014 Aug;21(4):174-80. doi: 10.3747/co.21.1984. PMID 25089099
- [Background] Pike CT, Birnbaum HG, Muehlenbein CE, Pohl GM, Natale RB. Healthcare costs and workloss burden of patients with chemotherapy-associated peripheral neuropathy in breast, ovarian, head and neck, and nonsmall cell lung cancer. Chemother Res Pract. 2012;2012:913848. doi: 10.1155/2012/913848. Epub 2012 Mar 14. PMID 22482054
- [Background] Lodewijckx J, Robijns J, Bensadoun RJ, Mebis J. Photobiomodulation Therapy for the Management of Chemotherapy-Induced Peripheral Neuropathy: An Overview. Photobiomodul Photomed Laser Surg. 2020 Jun;38(6):348-354. doi: 10.1089/photob.2019.4771. Epub 2020 May 28. PMID 32460667
- [Background] Rivera E, Cianfrocca M. Overview of neuropathy associated with taxanes for the treatment of metastatic breast cancer. Cancer Chemother Pharmacol. 2015 Apr;75(4):659-70. doi: 10.1007/s00280-014-2607-5. Epub 2015 Jan 18. PMID 25596818
- [Background] Li L, Huang Y, An C, Jing N, Xu C, Wang X, Li H, Tan T. Acupuncture in the treatment of chemotherapy-induced peripheral neuropathy: a meta-analysis and data mining. Front Neurol. 2024 Oct 29;15:1442841. doi: 10.3389/fneur.2024.1442841. eCollection 2024. PMID 39555482
- [Background] D'Souza RS, Her YF, Jin MY, Morsi M, Abd-Elsayed A. Neuromodulation Therapy for Chemotherapy-Induced Peripheral Neuropathy: A Systematic Review. Biomedicines. 2022 Aug 7;10(8):1909. doi: 10.3390/biomedicines10081909. PMID 36009456
- [Background] Brami C, Bao T, Deng G. Natural products and complementary therapies for chemotherapy-induced peripheral neuropathy: A systematic review. Crit Rev Oncol Hematol. 2016 Feb;98:325-34. doi: 10.1016/j.critrevonc.2015.11.014. Epub 2015 Nov 23. PMID 26652982
- [Background] Zhang X, Wang A, Wang M, Li G, Wei Q. Non-pharmacological therapy for chemotherapy-induced peripheral neurotoxicity: a network meta-analysis of randomized controlled trials. BMC Neurol. 2023 Dec 11;23(1):433. doi: 10.1186/s12883-023-03485-z. PMID 38082216
- [Background] Butkovic D, Toljan S, Matolic M, Kralik S, Radesic L. Comparison of laser acupuncture and metoclopramide in PONV prevention in children. Paediatr Anaesth. 2005 Jan;15(1):37-40. doi: 10.1111/j.1460-9592.2004.01388.x. PMID 15649161
- [Background] Gottschling S, Meyer S, Gribova I, Distler L, Berrang J, Gortner L, Graf N, Shamdeen GM. Laser acupuncture in children with headache: a double-blind, randomized, bicenter, placebo-controlled trial. Pain. 2008 Jul 15;137(2):405-412. doi: 10.1016/j.pain.2007.10.004. Epub 2007 Nov 19. PMID 18022318
- [Background] Klausner G, Troussier I, Canova CH, Bensadoun RJ. Clinical use of photobiomodulation as a supportive care during radiation therapy. Support Care Cancer. 2022 Jan;30(1):13-19. doi: 10.1007/s00520-021-06518-w. No abstract available. PMID 34623486
- [Background] de Pauli Paglioni M, Araujo ALD, Arboleda LPA, Palmier NR, Fonseca JM, Gomes-Silva W, Madrid-Troconis CC, Silveira FM, Martins MD, Faria KM, Ribeiro ACP, Brandao TB, Lopes MA, Leme AFP, Migliorati CA, Santos-Silva AR. Tumor safety and side effects of photobiomodulation therapy used for prevention and management of cancer treatment toxicities. A systematic review. Oral Oncol. 2019 Jun;93:21-28. doi: 10.1016/j.oraloncology.2019.04.004. Epub 2019 Apr 10. PMID 31109692
- [Background] Chung H, Dai T, Sharma SK, Huang YY, Carroll JD, Hamblin MR. The nuts and bolts of low-level laser (light) therapy. Ann Biomed Eng. 2012 Feb;40(2):516-33. doi: 10.1007/s10439-011-0454-7. Epub 2011 Nov 2. PMID 22045511
- [Background] Bjordal JM, Couppe C, Chow RT, Tuner J, Ljunggren EA. A systematic review of low level laser therapy with location-specific doses for pain from chronic joint disorders. Aust J Physiother. 2003;49(2):107-16. doi: 10.1016/s0004-9514(14)60127-6. PMID 12775206
- [Background] Khamseh ME, Kazemikho N, Aghili R, Forough B, Lajevardi M, Hashem Dabaghian F, Goushegir A, Malek M. Diabetic distal symmetric polyneuropathy: effect of low-intensity laser therapy. Lasers Med Sci. 2011 Nov;26(6):831-5. doi: 10.1007/s10103-011-0977-z. Epub 2011 Aug 19. PMID 21853320
- [Background] Cg SK, Maiya AG, Hande HM, Vidyasagar S, Rao K, Rajagopal KV. Efficacy of low level laser therapy on painful diabetic peripheral neuropathy. Laser Ther. 2015 Oct 2;24(3):195-200. doi: 10.5978/islsm.15-OR-12. PMID 26557734
- [Background] Hsieh YL, Chou LW, Hong SF, Chang FC, Tseng SW, Huang CC, Yang CH, Yang CC, Chiu WF. Laser acupuncture attenuates oxaliplatin-induced peripheral neuropathy in patients with gastrointestinal cancer: a pilot prospective cohort study. Acupunct Med. 2016 Oct;34(5):398-405. doi: 10.1136/acupmed-2016-011112. Epub 2016 Sep 9. PMID 27613370
- [Background] Pereira FC, Parisi JR, Maglioni CB, Machado GB, Barragan-Iglesias P, Silva JRT, Silva ML. Antinociceptive effects of low-level laser therapy at 3 and 8 j/cm2 in a rat model of postoperative pain: possible role of endogenous Opioids. Lasers Surg Med. 2017 Nov;49(9):844-851. doi: 10.1002/lsm.22696. Epub 2017 Jul 3. PMID 28671718
- [Background] Wang CZ, Chen YJ, Wang YH, Yeh ML, Huang MH, Ho ML, Liang JI, Chen CH. Low-level laser irradiation improves functional recovery and nerve regeneration in sciatic nerve crush rat injury model. PLoS One. 2014 Aug 13;9(8):e103348. doi: 10.1371/journal.pone.0103348. eCollection 2014. PMID 25119457
- [Background] Hsieh YL, Fan YC, Yang CC. Low-level laser therapy alleviates mechanical and cold allodynia induced by oxaliplatin administration in rats. Support Care Cancer. 2016 Jan;24(1):233-242. doi: 10.1007/s00520-015-2773-y. Epub 2015 May 26. PMID 26006084
- [Background] Argenta PA, Ballman KV, Geller MA, Carson LF, Ghebre R, Mullany SA, Teoh DG, Winterhoff BJ, Rivard CL, Erickson BK. The effect of photobiomodulation on chemotherapy-induced peripheral neuropathy: A randomized, sham-controlled clinical trial. Gynecol Oncol. 2017 Jan;144(1):159-166. doi: 10.1016/j.ygyno.2016.11.013. Epub 2016 Nov 22. PMID 27887804
- [Background] Marcus J, Lasch K, Wan Y, Yang M, Hsu C, Merante D. An Assessment of Clinically Important Differences on the Worst Pain Severity Item of the Modified Brief Pain Inventory in Patients with Diabetic Peripheral Neuropathic Pain. Pain Res Manag. 2018 Jul 22;2018:2140420. doi: 10.1155/2018/2140420. eCollection 2018. PMID 30140328
- [Background] Cleeland CS, Ryan KM. Pain assessment: global use of the Brief Pain Inventory. Ann Acad Med Singap. 1994 Mar;23(2):129-38. PMID 8080219
- [Background] Poundja J, Fikretoglu D, Guay S, Brunet A. Validation of the French version of the brief pain inventory in Canadian veterans suffering from traumatic stress. J Pain Symptom Manage. 2007 Jun;33(6):720-6. doi: 10.1016/j.jpainsymman.2006.09.031. PMID 17531912
- [Background] Atkinson TM, Mendoza TR, Sit L, Passik S, Scher HI, Cleeland C, Basch E. The Brief Pain Inventory and its "pain at its worst in the last 24 hours" item: clinical trial endpoint considerations. Pain Med. 2010 Mar;11(3):337-46. doi: 10.1111/j.1526-4637.2009.00774.x. Epub 2010 Jan 15. PMID 20030743
- [Background] Bouhassira D. Neuropathic pain: Definition, assessment and epidemiology. Rev Neurol (Paris). 2019 Jan-Feb;175(1-2):16-25. doi: 10.1016/j.neurol.2018.09.016. Epub 2018 Oct 29. PMID 30385075
- [Background] Bouhassira D, Luporsi E, Krakowski I. Prevalence and incidence of chronic pain with or without neuropathic characteristics in patients with cancer. Pain. 2017 Jun;158(6):1118-1125. doi: 10.1097/j.pain.0000000000000895. PMID 28267066
- [Background] Bouhassira D, Attal N, Fermanian J, Alchaar H, Gautron M, Masquelier E, Rostaing S, Lanteri-Minet M, Collin E, Grisart J, Boureau F. Development and validation of the Neuropathic Pain Symptom Inventory. Pain. 2004 Apr;108(3):248-257. doi: 10.1016/j.pain.2003.12.024. PMID 15030944
- [Background] Hawker GA, Mian S, Kendzerska T, French M. Measures of adult pain: Visual Analog Scale for Pain (VAS Pain), Numeric Rating Scale for Pain (NRS Pain), McGill Pain Questionnaire (MPQ), Short-Form McGill Pain Questionnaire (SF-MPQ), Chronic Pain Grade Scale (CPGS), Short Form-36 Bodily Pain Scale (SF-36 BPS), and Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S240-52. doi: 10.1002/acr.20543. No abstract available. PMID 22588748
- [Background] Calhoun EA, Welshman EE, Chang CH, Lurain JR, Fishman DA, Hunt TL, Cella D. Psychometric evaluation of the Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity (Fact/GOG-Ntx) questionnaire for patients receiving systemic chemotherapy. Int J Gynecol Cancer. 2003 Nov-Dec;13(6):741-8. doi: 10.1111/j.1525-1438.2003.13603.x. PMID 14675309
- [Background] Conroy T, Mercier M, Bonneterre J, Luporsi E, Lefebvre JL, Lapeyre M, Puyraveau M, Schraub S. French version of FACT-G: validation and comparison with other cancer-specific instruments. Eur J Cancer. 2004 Oct;40(15):2243-52. doi: 10.1016/j.ejca.2004.06.010. PMID 15454249
- [Background] Savard MH, Savard J, Simard S, Ivers H. Empirical validation of the Insomnia Severity Index in cancer patients. Psychooncology. 2005 Jun;14(6):429-41. doi: 10.1002/pon.860. PMID 15376284
- [Background] Bayard S, Madiouni C, Niel Carlos C, Cornu C, Moulin A, Raffard S. French adult normative data for a Standard Executive Neuropsychological Test Battery. Arch Clin Neuropsychol. 2025 Apr 27;40(3):486-497. doi: 10.1093/arclin/acad062. PMID 37565605